CLINICAL TRIAL: NCT06177028
Title: MCLENA-2: A Phase II Clinical Trial for the Assessment of Biomarker Trajectory in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease Treated With Lenalidomide (Amendment to IND # 142121)
Brief Title: MCLENA-2: A Phase II Clinical Trial for the Assessment of Lenalidomide in Patients With Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013717
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Impairment, Mild; Cognitive Dysfunction; Amyloid Plaque; Neurodegenerative Disease, Hereditary; Inflammation, Brain
Keywords: Alzheimer's disease; CSF; Biomarkers; Brain Imaging; Brain Amyloid; Memory Loss; Immunomodulation
MeSH Terms: conditions — Cognitive Dysfunction; Plaque, Amyloid; Heredodegenerative Disorders, Nervous System; Encephalitis; Alzheimer Disease; Memory Disorders | interventions — Lenalidomide

STUDY DESIGN:
Intervention Model Description: This study will take place at a single site. We will enroll 45 male and female participants, 50-90 years of age, in general good health, with mild cognitive impairment due to AD. The trial will last up to 30 weeks in duration. Lenalidomide 10 mg/day vs. placebo taken daily orally (ratio 2:1).
  Participants completing the study will be involved for up to 45 weeks in duration, from screening to end of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Beside the clinical pharmacologist and biostatistician, all parties involved in the present study will be blinded until all data are collected, including medical staff, patients and his/her car giver, imaging staff, and scientists collecting data from biosamples. The blinding will be lifted only after all data are acquired, and before statistical analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lenalidomide (Experimental): Lenalidomide 10 mg/day taken daily orally for 26 weeks of treatment followed by 4 weeks of washout. The trial will last up to 30 weeks in duration.
  Interventions: Drug: Lenalidomide 10 mg
- Placebo (Placebo Comparator): Placebo taken daily orally for 26 weeks of treatment followed by 4 weeks of washout. The trial will last up to 30 weeks in duration.
  Interventions: Drug: Lenalidomide 10 mg

INTERVENTIONS:
Drug: Lenalidomide 10 mg — Lenalidomide is a cancer drug, It is also known by it's brand name Revlimid.
  Other Names: Lenalid

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel group study. The use of placebo is appropriate to minimize bias related to treatment expectations of the subject, study partner, and site investigator, as well as to changes in the relationship between the subject and study partner that might occur with the initiation of treatment and expectation of improvement in motor symptoms or cognition. Changes in subject/study partner interactions can impact subject mood and might introduce biases that cannot be quantified. The double-blind use of placebo will also prevent bias in the clinical and scientific assessments.

DETAILED DESCRIPTION:
There are currently no FDA-approved medications indicated for the treatment of AD. While inflammation is pervasive to many neurological disorders, no clinical trial has yet demonstrated the efficacy of anti-inflammatory agents for AD. Interestingly, chronic peripheral low-grade inflammation is associated with aging and increases the risk for disease and mortality, including AD. Accumulating evidence indicates that nuclear factor-kappa B, tumor necrosis factor alpha (TNFα), interleukins (e.g. IL-1beta, IL-2, and IL-6), and chemokines (e.g. IL-8) are found elevated both in the blood and central nervous system (CNS) of AD patients. These data confirm that inflammation plays a central role in the cause and effect of AD neuropathology.

The immunomodulator, anti-cancer agent lenalidomide is one of the very few pleiotropic agents that both lowers the expression of TNFα, IL-6, IL-8, and increases the expression of anti-inflammatory cytokines (e.g. IL-10), to modulate both innate and adaptive immune responses. In the current project we aim to test the central hypothesis that lenalidomide reduces inflammatory and AD-associated pathological biomarkers in the blood and CSF. For this, we designed a 6-month, Phase II, double blind, randomized, two-armed, parallel group, placebo controlled, and proof-of-mechanism clinical study in early symptomatic AD subjects (i.e. amnestic mild cognitive impairment; aMCI). The effects of lenalidomide treatment will be assessed continuously for 26 weeks and 4 weeks washout (total of 30 weeks).

ELIGIBILITY:
In order to be eligible for this study, subjects must meet the following inclusion criteria:

Inclusion Criteria:

1. Male or female outpatients.
2. At least 50 years of age, but less than 90 (89 at time of screening)
3. Females must be surgically sterile (bilateral tubal ligation, oophorectomy, or hysterectomy) or postmenopausal for 2 years (no women at risk of pregnancy will be accepted in this study).
4. Must have been diagnosed with amnestic MCI based on the most recent NIA-AA criteria (Albert et al., 2011), i.e. at both the screening and baseline visits (visits 1 and 2) have a documented Mini Mental State Exam (MMSE) score between 22-28.
5. CT or MRI scan of the brain obtained during the course of the dementia must be consistent with the diagnosis and show no evidence of significant focal lesions or of pathology which could contribute to dementia. If neither a CT nor an MRI scan is available from the past 12 months, a CT scan fulfilling the requirements must be obtained before randomization.
6. Vision and hearing must be sufficient to comply with study procedures.
7. Be able to take oral medications.
8. Hachinski ischemic score must be ≤ 4.
9. Geriatric depression scale must be ≤ 10.
10. Can be on stable doses of a cholinesterase inhibitor and/or memantine as long as it is stable for at least 90 days before screening and is expected to remain on a stable dose for the remainder of the study period; or have demonstrated intolerance to or lack of efficacy from these medications.
11. Must have a collateral informant/study partner who has significant direct contact with the patient at least 10 hours per week and who is willing to accompany the patient to specified clinic visits, supervise administration of all study medication, and be available for telephone visits/interviews.
12. If the patient has a legally authorized representative (LAR), the LAR must review and sign the informed consent form. If the patient does not have an LAR, the patient must appear able to provide informed consent and must review and sign the informed consent form. In addition, the patient's informant/study partner (as defined above) must sign an informed consent form. If the LAR and the patient's informant /study partner is the same individual, he/she should sign under both designations.
13. Must reside in the community.
14. Patients with stable prostate cancer may be included at the discretion of the Medical Monitor.
15. Positivity for amyloid brain scan: Amyloid PET positive at SUVr of 1.05

Exclusion Criteria:

Subjects will be excluded if they have any of the condition listed below:

1. Current evidence or history within the last 3 years of a neurological or psychiatric illness that could contribute to dementia, including (but not limited to) epilepsy, focal brain lesion, Parkinson's disease, seizure disorder, head injury with loss of consciousness
2. DSM IV criteria for any major psychiatric disorder including psychosis, major depression and bipolar disorder.
3. Unwilling or unable to undergo a Lumbar Puncture.
4. Known history or self-reported alcohol or substance abuse.
5. Living alone.
6. Poorly controlled hypertension. 7 .History of myocardial infarction or signs or symptoms of unstable coronary artery disease within the last year (including revascularization procedure/angioplasty).

8. Severe pulmonary disease (including chronic obstructive pulmonary disease) requiring more than 2 hospitalizations within the past year.

9. Untreated sleep apnea. 10. Any thyroid disease (unless euthyroid on treatment for at least 6 months prior to screening).

11. Active neoplastic disease (except for skin tumors other than melanoma) within five years.

12. History of multiple myeloma. 13. Absolute neutropenia of <750/mm3, or a history of neutropenia. 14. History of or current thromboembolism (including deep venous thrombosis). 15. Any clinically significant hepatic or renal disease (including presence of Hepatitis B or C antigen/antibody or an elevated transaminase levels of greater than two times the upper limit of normal (ULN) or creatinine greater than 1.5 x ULN).

16. Clinically significant hematologic or coagulation disorder including any unexplained anemia or a platelet count less than 100,000/μL at screening.

17. Use of any investigational drug within 30 days or within five half-lives of the investigational agent, whichever is longer.

18. Use any investigational medical device within two weeks before screening or after end of the present study.

19. Females who are at risk of pregnancy or are of child bearing age. 20. Unwilling or unable to undergo MRI and PET imaging. 21. Cardiac pacemaker or defibrillator or other implanted device. 22. In the opinion of the investigator, participation would not be in the best interest of the subject

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-01-02 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of lenalidomide | After 26 weeks of treatment
  To assess the effect of lenalidomide on inflammatory markers in CSF and blood, as well as safety and toxicity.

SECONDARY OUTCOMES:
To asses the effect of lenalidomide | 26 weeks of treatment
  : To assess the effects of lenalidomide on CSF makers of AD (e.g. amyloid beta and tau levels) in aMCI patients

IPD SHARING:
Plan to Share IPD: Yes
The protocol used and data collected in the course of this study will be shared with other researchers. The protocol will be published in a scientific journal and presented as posters in scientific meetings. Data and remaining bio samples, after deidentification, will be made available to the community 6 months after publication of the results of the study in peer-reviewed articles.
Supporting Information: Study Protocol
Access Criteria: Papers will be accessible online Data and bio samples can be requested from the principal investigator 6 months after publication of the results of the study in peer-reviewed articles